CLINICAL TRIAL: NCT06796790
Title: Efficacy and Mechanisms of Media and Storybook Interventions to Promote Children's Early Literacy Skills Via Caregiver Engagement
Brief Title: Literacy Instruction Through Media for Everyone
Acronym: LIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Central Florida (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rebecca Dore, Director of Research, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AWD - 118236; R01HD114687 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Media Effects on Literacy Gains in Young Children
Keywords: Literacy; Media; Shared reading; Poverty; Parents; Intervention; Preschool; Television
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial hybrid type 2 design with three planned variations: (1) caregiver-led media-based early literacy intervention, (2) caregiver-led shared reading early literacy intervention, and (3) business-as-usual control. Literacy based media and shared reading will be used that promote literacy learning. Families enrolled in groups (1) and (2) will complete 12 weeks intervention. Families in all groups will also have follow ups at 3-, 6-, and 12-months post-intervention to test long-term effects. Families will digitally log their intervention sessions to track adherence as well as audio record 1 weekly session. Caregivers will be surveyed pre-intervention on other family characteristics and children will be assessed at pre-intervention, post-intervention, 3-, 6-, and 12-months post-intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Media instruction (Experimental): Caregivers will be asked to implement joint media sessions with their child four times per week for 12 weeks using lightly adapted versions of the commercially-available Super Why! program, which focuses on early literacy skills, including alphabet knowledge, rhyming, spelling, and print concepts. Sessions are anticipated to last 20 minutes. Caregivers will be trained by researchers on explicit strategies to use to promote children's learning. Caregivers will digitally log every session and audio record 1 session each week.
  Interventions: Behavioral: Media instruction
- Storybook instruction (Active Comparator): Caregivers will be asked to implement joint storybook reading sessions with their child four times per week for 12 weeks using adapted versions of the commercially -available Super-Why! storybooks, which focus on early literacy skills including alphabet knowledge, rhyming, spelling, and print concepts. Sessions are anticipated to last 20 minutes. Caregivers will be trained by researchers on explicit strategies to use to promote children's learning. Caregivers will digitally log every session and audio record 1 session each week.
  Interventions: Behavioral: Storybook intervention
- Business-as-usual control (No Intervention): Caregivers will be asked to log any joint learning activities they engage in with their child but will not be provided with any specific materials or instructions.

INTERVENTIONS:
Behavioral: Media instruction — Caregivers will be asked to implement joint media sessions with their child four times per week for 12 weeks using lightly adapted versions of the commercially-available Super Why! program, which focuses on early literacy skills, including alphabet knowledge, rhyming, spelling, and print concepts. Sessions are anticipated to last 20 minutes. Caregivers will be trained by researchers on explicit strategies to use to promote children's learning. Caregivers will digitally log every session and audio record 1 session each week
  Arms: Media instruction
Behavioral: Storybook intervention — Caregivers will be asked to implement joint storybook reading sessions with their child four times per week for 12 weeks using adapted versions of the commercially -available Super-Why! storybooks, which focus on early literacy skills including alphabet knowledge, rhyming, spelling, and print concepts. Sessions are anticipated to last 20 minutes. Caregivers will be trained by researchers on explicit strategies to use to promote children's learning. Caregivers will digitally log every session and audio record 1 session each week.
  Arms: Storybook instruction

SUMMARY:
The goal of this study is to determine whether an intervention to support caregivers in engaging with their children while using educational media together can improve children's early literacy skills, compared to an aligned shared book reading intervention and to no intervention. Given that early literacy skills predict children's later academic learning, this home intervention, which aims to shape the communication patterns surrounding a common, family-friendly activity, has the potential to positively influence the trajectory of low income children's academic success. The investigators propose that amedia based activity will reduce barriers and increase adherence therefore increasing literacy skills over time.

DETAILED DESCRIPTION:
The proposed study draws upon an implementation science framework (Nilsen, 2015) to determine the extent to which a media-based caregiver-led intervention improves caregiver adherence and in turn children's early literacy development relative to a shared reading intervention. Caregiver-implemented shared reading interventions represent the 'current standard practice' for addressing early literacy needs, yet many caregivers cannot implement this practice with adequate adherence. This is particularly true for low-socioeconomic status families, in which shared reading may not be a conventional activity and barriers inhibit its use. The investigators propose-and test-that a media-based intervention reduces barriers to intervention implementation and increases social validity, leading to higher levels of adherence and, via mediation, enhanced child literacy outcomes. To establish this causal chain, the investigators mplement a media-based early literacy intervention, compare it to a highly aligned shared reading intervention, and measure (1) social validity of the intervention to test whether use of media circumvents barriers, (2) caregiver adherence (i.e., frequency and dosage), and (3) child early literacy skills gains immediately and over time. As the first causally interpretable study to compare media and shared reading as caregiver-led interventions, the proposed project will identify strategies to improve adherence in home-based interventions and inform development of interventions to improve school readiness among low-SES children.

ELIGIBILITY:
Inclusion Criteria:

* between 42 and 57 months at enrollment
* minimally verbal in English
* caregiver sufficiently proficient in English
* does not have severe intellectual disability

Exclusion Criteria:

* under 42 months
* over 57 months at enrollment
* severe intellectual disability
* not proficient in English

Ages: 42 Months to 57 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Print concept knowledge | At pretest after enrollment and at posttest after the 12 week intervention period
  Children are administered the Preschool Word and Print Awareness (PWPA) measure (Justice et al., 2006), which examines children's knowledge of 16 basic print concepts. The PWPA has high inter-rater reliability (96% to 100%, Justice & Ezell, 200), acceptable internal consistency (#= .7; Dobbs- Oates et al., 2015) and can reliably estimate preschoolers' print-concept knowledge (Justice et al., 2006).
Alphabet knowledge | At pretest after enrollment and at posttest after the 12 week intervention period
  Children are administered the Alphabet Knowledge subtest of the Phonological Awareness Literacy Screening - Preschool (PALS-PreK; Invernizzi et al., 2001). Children are presented with uppercase and lowercase letters printed in random order and receive a point for each letter named correctly.
  Cronbach's alphas average average .86. Inter-rater reliability is >.96 (Invernizzi et al., 2004). The full PALS-PreK test is highly correlated with measures of reading ability (e.g., Test of Early Reading Ability, r= .67) and predicts later performance on a similar literacy measure (rs > .53). Further, this subtest has high predictive validity in discriminating children who will later be identified as needing additional instruction (Invernizzi et al., 2001).
Name Writing | At pretest after enrollment and at posttest after the 12 week intervention period
  Children are administered the Name Writing subtest from the PALS-PreK. In the Name Writing subtest, the child is asked to draw a picture of themselves and then write their name. They are then asked to show the assessor their name. Only the written name is scored. This subtests has high inter-rater reliability (.99). As noted above, the full test has good convergent and predictive validity (Invernizzi et al., 2001).
Phonological Awareness | At pretest after enrollment and at posttest after the 12 week intervention period
  Children are administered two subtests from the PALS-PreK. In the Beginning Sound Awareness subtest, the child is asked to produce the beginning sound of a word. In the Rhyme Awareness subtest, the experimenter says a word and asks the child to point to the picture that rhymes. These subtests have acceptable reliability (# = .93 and # = .84) and inter-rater reliability is high (.99). As noted above, the full test has good convergent and predictive validity (Invernizzi et al., 2001).
Word reading | At pretest after enrollment, at posttest after the 12 week intervention period, at 3-month follow up, at 6-month follow-up, and at 12- month follow up
  At all timepoints, children are administered the Letter-Word Identification subtest of the Woodcock Johnson IV Test of Achievement (WJ IV; Schrank, McGrew & Mather, 2014). This subtest requires children to identify or read isolated letters and words orally. This subtest has adequate internal-consistency (.94; Schrank & Wendling, 2018). It has a high factor loading onto the Broad Reading cluster (.92; McGrew et al., 2014) which is highly correlated with other measures of reading like the Wechsler Individual Achievement Test (WIAT) Total Reading (.89; Schrank & Wendling, 2018). It is strongly correlated with general school readiness (r = .84) as measured by the Differential Ability Scales (McGrew et al., 2014).
Spelling | At pretest after enrollment, at posttest after the 12 week intervention period, at 3-month follow up, at 6-month follow-up, and at 12- month follow up
  At all timepoints, children are administered the Spelling subtest from the WJ IV, requiring children to draw lines, trace and write letters, and spell orally presented words. This subtest has adequate internal-consistency reliability (.92; Schrank & Wendling, 2018) and a high factor loading onto the Broad Written Language Cluster (.87), which is highly correlated with other measures of writing like WIAT Written Expression (.77; McGrew et al., 2014). This subtest is moderately correlated (r = .69) with general school readiness as measured by the Differential Ability Scales (McGrew et al., 2014).

SECONDARY OUTCOMES:
Enjoyment of intervention activities | Four times per week during the 12-week intervention and at posttest after the intervention
  Enjoyment of intervention activities is measured to assess the extent to which the media intervention circumvents barriers related to caregiver difficulty and discomfort with reading. Enjoyment will be measured with three items: "How do you think today's session went?", "How much did you enjoy these sessions?", and "How uncomfortable or difficult did you find these sessions?"
Perceived value of intervention activities | At posttest after the 12 week intervention period
  Perceived value of intervention activities is measured to assess the extent to which the media intervention reduces barriers related to a limited understanding of the benefits of shared-reading activities. Two items are used: "How much did these sessions help your child's development?" and "How much did these sessions help your child learn about letters and how to read simple words?".
Ease of Scheduling | At posttest after the 12 week intervention period
  Ease of fitting activities into schedule is measured to assess the extent to which the media intervention reduces the time pressure barrier. One item asks: "How easy was it to fit this session into your family's schedule?"
Caregiver Adherence | Throughout the 12-week intervention
  Caregivers will be trained in procedures for using a digital Qualtrics log to track use of the intervention activities. The log will be preloaded as a bookmark onto the home screen of each tablet and will ask participants to note the episode watched.
Quantity of print-related talk | Throughout the 12-week intervention
  Audio-recorded intervention sessions will be coded by trained research staff to document the quantity of print-related talk within each session. Specifically, the Fidelity Coding Catalog (FCC) coding scheme was developed to document caregiver-child talk during reading sessions and is a reliable event-based coding system measuring frequency and quantity of print-focused talk. The FCC captures, for instance, every adult utterance that contains print-related key words, such as letter, word, and read. The quantity of print-related talk as measured by the FCC is an important index of intervention adherence but also represents a key mechanism through which intervention impacts early literacy development (McGinty et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Dore, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Crane Center for Early Childhood, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate quantitative data from 450 families and children, which will be used to assess the efficacy of a media-based early literacy intervention. The data will be collected via direct assessments, questionnaires, applications loaded onto provided tablets, and audio and video observations. The primary final, cleaned data will consist of a single comma-delimited file for all valid responses. Transcription records will be stored as text files and audio/video files will be stored as MP3/4 files. Upon publication of major findings from the proposed study, the primary data file, transcripts, and audio and video files will be shared with other researchers through the Open Science Framework (primary comma-delimited data file), Databrary (audio and video files), and CHILDES/TalkBank (transcripts).
Time Frame: Data will be made available upon publication of major findings from the proposed study. Study data deposited in the OSF, Databrary, and CHILDES/TalkBank will be available to the research community in perpetuity.
Access Criteria: Deidentified datasets will be made available as public use data on the OSF. Data with potentially personally identifiable information, such as audio or video, will be shared in more restricted manner via Databrary. Databrary provides data access to authorized users who have been granted secure access by Databrary's administrators. Only researchers with Principal Investigator status from institutions with Institutional Review Boards or similar review entities, or researchers affiliated with Principal Investigators, will be authorized for access. Transcripts will be shared via CHILDES/TalkBank and will be redacted as needed to remove potentially personally identifiable information.